CLINICAL TRIAL: NCT07065643
Title: GendAge Weight Loss Study: Sex Hormones as Regulators of the Age- and Sex-dependent Benefits of Caloric Restriction
Brief Title: Sex Hormones as Regulators of the Age- and Sex-dependent Benefits of Caloric Restriction
Acronym: GendAge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 822; 2-034-25 (Other Grant/Funding Number: Medical Research Council (MRC))
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Overweight and Obese Adults; Healthy
Keywords: caloric restriction; low calorie diet; menopause; overweight; obesity; weigh loss; ageing; energy expenditure; body composition
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Young women (Experimental): Age: 18 to 40 years old
  Interventions: Other: Phase 1 - Maintenance Diet; Other: Phase 2 - Weight loss diet
- Young men (Active Comparator): Age: 18 to 40 years old
  Interventions: Other: Phase 1 - Maintenance Diet; Other: Phase 2 - Weight loss diet
- Older women (menopause & no-HRT) (Experimental): Age 55-65 years, in menopause, not taking Hormonal Replacement Therapy (HRT)
  Interventions: Other: Phase 1 - Maintenance Diet; Other: Phase 2 - Weight loss diet
- Older women (menopause & HRT) (Experimental): Age 55-65 years, in menopause, who have continuously taken oestrogen HRT for 24 months
  Interventions: Other: Phase 1 - Maintenance Diet; Other: Phase 2 - Weight loss diet
- Older men (Active Comparator): Age 55-65 years
  Interventions: Other: Phase 1 - Maintenance Diet; Other: Phase 2 - Weight loss diet

INTERVENTIONS:
Other: Phase 1 - Maintenance Diet — 3d maintenance diet (MT, fixed macronutrient composition of 15% protein, 30% fat and 55% CHO), fed to energy requirements (1.3 X RMR)
Other: Phase 2 - Weight loss diet — 6 week calorie restricted high protein diet (CR, fixed macronutrient composition as 30% protein, 35% fat and 35% CHO) fed to energy requirements [0.8 X Resting Metabolic Rate (RMR)], with stepwise reduction of 100kcal/d at week 3 and 5

SUMMARY:
Obesity increases the risk of type 2 diabetes, cardiovascular disease, and certain cancers, primarily due to elevated abdominal fat storage. With nearly two-thirds of the UK population living with overweight or obesity, there is an urgent necessity for evidence-based public health guidance to promote healthy weight. Calorie deficit can facilitate weight loss and body fat reduction, leading to health benefits, such as improved blood glucose control. Current weight management advice centres on lifestyle modification, incorporating changes to diet and physical activity to support a calorie deficit. However, existing dieting recommendations fail to consider gender or age. This is a surprising oversight, as it is well established that health outcomes vary significantly between men and women across the lifespan. Further, the menopause may have an impact on fat storage linked to changes in sex hormones. Our recent research, involving both mice and humans, has indicated that females are less responsive to weight loss and fat reduction during dieting. This study aims to understand endocrine and metabolic sex-based differences in obesity and calorie restriction, with a particular focus on women's health. We plan to conduct a diet study with 75 participants, encompassing both younger and older men and women, to monitor changes in energy expenditure and body composition using gold-standard techniques, such as doubly-labelled water. Blood and abdominal fat tissue samples will be collected to investigate how sex hormones might elucidate these differences. The aim of the study is to enhance our understanding of diet and women's health to combat obesity and promote healthy ageing.

ELIGIBILITY:
Inclusion criteria

* Adults (aged over 18years) who are healthy but overweight/obese (BMI 27-45kg/m2) males and females as:
* 15 women (age 40 or less years)
* 15 men (age 40 or less years)
* 15 women (age 55-65 years) in menopause*; not taking Hormone Replacement Therapy (HRT)
* 15 men (age 55-65 years)
* 15 women (age 55-65 years) in menopause; taking HRT**

  * menopause definition is no menstrual period for 12 months **HRT inclusion criteria - women will have continuously taken oestrogen HRT for 24 months

Exclusion criteria:

Potential volunteers will be asked to fill in a health questionnaire at the screening visit to assess their suitability for the study. This information will allow us to exclude participants.

Medication exclusion criteria, current use :-

• weight loss medication (e.g. GLP agonists), β-blockers, antihistamines, antipsychotics, benzodiazepines, barbiturates, melatonin, Ritalin, modafinil, soporifics, hypnotics, antiepileptic drugs, diabetes medication (e.g. metformin or insulin).

Self-reported medical exclusion criteria:

* Females who are planning to be pregnant, are pregnant or are breastfeeding
* Anyone with coeliac disease or gluten intolerance or food allergy
* Anyone with diagnosed T1 or T2 diabetes
* Anyone suffering from a psychiatric disorder or any type of substance abuse

Other exclusion criteria

* Anyone following a vegetarian or vegan diet
* Anyone currently following a weight loss programme (that may be affecting lifestyle, physical activity & diet) or undergone gastric band/reduction surgery; including GLP agonist (e.g. Semaglutide injection, Ozempic®).
* Anyone currently participating in another research study
* Anyone with unsuitable veins for blood sampling
* Anyone who is unable to fluently speak, read and understand English
* Anyone who is unable to comply to an alcohol-free diet for 6 weeks
* Anyone unable to give fully informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biological (cisgender) males and females
Enrollment: 75 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in body mass expressed as weight in kilograms (kg) | From baseline (day 1) to end of intervention (day 53); additional measurements taken three times a week throughout the intervention duration
  Measured using digital scale
Change in energy expenditure expressed in kilocalories per day (kcal/day) | From day 11 (start of the calorie-restricted diet) to the end of the intervention (day 52); with additional doses consumed on day 25 and 39
  Measured using stable isotope method - doubly labelled water (DLW) - with urine sample collection

SECONDARY OUTCOMES:
Change in resting metabolic rate (RMR) expressed in kcal/day | From day 8 (start of the maintenance diet) to end of the intervention (day 53)
  Measured using ventilated hood indirect calorimetry
Change in bone mineral content in grams (g) | From day 8 (start of the maintenance diet) to end of the intervention (day 53)
  Measured using Dual Energy X-Ray Absorptiometry (DXA) scan
Change in total body water (TBW) in litres (l) | From day 11 (start of the calorie-restricted diet) to end of the intervention (day 53)
  Measured using deuterium dilution, with urine sample collection
Change in total body density expressed in litres (l) | From day 8 (start of the maintenance diet) to end of the intervention (day 53)
  Measured using BodPod air displacement plethysmography
Change in body fat-mass percentage (%) | From day 8 (start of the maintenance diet) to end of the intervention (day 53)
  Derived from Lohman's 4-compartment model (body mass; body density; total body water; and bone mineral content)
Change in non-esterified fatty acids (NEFA) concentration in fasted blood sample | From day 8 (start of the maintenance diet) to end of the intervention (day 53); also measured at midpoint of calorie-restricted diet (day 32)
  Analysed by KONE
Change in concentration of caloric-restriction (CR) related hormones in fasted blood sample | From day 8 (start of the maintenance diet) to end of the intervention (day 53); also measured at midpoint of calorie restricted diet (day 32)
  Includes: leptin, adiponectin, cortisol; analysed by ELISA
Change in sex hormones concentration in fasted blood sample | From day 8 (start of the maintenance diet) to end of the intervention (day 53); also measured at midpoint of calorie restricted diet (day 32)
  Includes: oestrogens, progesterone, androgens; analysed by high -sensitivity liquid chromatography-mass spectrometry (LC-MS)
Body height measured in meters (m) | Only at baseline
  Measured using stadiometer
Change in Body Mass Index (BMI) expressed as kg/m^2 | From baseline (day 1) to end of intervention (day 53); additional measurements taken three times a week throughout the intervention duration
  BMI will be calculated using weight and height measures
Change in adipose tissue metabolism assessed by adipocite size | From day 8 (start of the maintenance diet) to end of the intervention (day 53)
  Measured via abdominal subcutaneous fat biopsy using fine needle aspiration and histomorphometry method
Change in adipose tissue metabolism assessed by phosphorylation of hormone-sensitive lipase (HSL) | From day 8 (start of the maintenance diet) to end of the intervention (day 53)
  Measured via abdominal subcutaneous fat biopsy using fine needle aspiration and immunoblotting method.

OTHER OUTCOMES:
Change in glycaemic control in response to caloric restriction diet | Every day of the study (days 1-53)
  Measured with continuous glucose monitoring (CGM) Freestyle Libre
Change in fasting concentration of glucose | From day 8 (start of the maintenance diet) to end of the intervention (day 53)
  Measured from capillary blood from a finger
Change in fasting concentration of ketones | From day 8 (start of the maintenance diet) to end of the intervention (day 53)
  Measured from capillary blood from a finger
Change in fasting concentration of Glucose Ketone Index (GKI) | From day 8 (start of the maintenance diet) to end of the intervention (day 53)
  Calculated from glucose and ketone values
Change in levels of physical activity (PA) expressed as energy expenditure (kcal/day) | Every day of the study (days 1-53)
  Actigraph wearable device for recording physical activity via accelerometery method
Change in physical activity intensity expressed as minutes spent on Moderate to vigorous (MVPA) per day | Every day of the study (days 1-53)
  Measured accelerometry (with Actigraph wearable device) and calculated using energy expenditure and time spent in MVPA
Change in food intake | Starting from ad libitum intake (days 1-7) and every day of the study diets (day 8-52)
  Measured using weighted intake record

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra M Johnstone, Professor, Principal Investigator — Rowett Institute, University of Aberdeen
Locations (1):
- Rowett Institute, University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The study will be registered with ClinicalTrials.gov as a data repository. Links to IPD that underlie results in publications will be made available at the appropriate time through the project team's website which will contain a summary of the data compiled.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be shared with the academic community once this has been published in open access journals
Access Criteria: Open access from the project's website to IPD that underline the results reported in scientific publications.

REFERENCES:
- See also: Project website — https://www.abdn.ac.uk/rowett/volunteer/current-studies/gendage-study/